CLINICAL TRIAL: NCT06299865
Title: Comparison of Detection Rates of Osteoporosis Between Dual Energy X-ray and Quantitative CT
Brief Title: Comparison of Detection Rates Between Two Commonly Used Bone Density Measurement Methods
Status: Not yet recruiting | Type: Observational
Sponsor: Xiaoqian Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaoqian Zhang, chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023（150）
Record Dates: First submitted 2024-01-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Osteoporosis; Diagnosis; Dual Energy X-ray Absorptiometry; Quantitative Computed Tomography
MeSH Terms: conditions — Osteoporosis; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ungrouped — Ungrouped

SUMMARY:
72 adult patients who underwent lumbar spine anteroposterior DXA and QCT examinations at Qianfoshan Hospital in Shandong Province from January 2019 to December 2022 were selected, with an interval of no more than 3 months between the two examinations for the same patient.

1. Record the patient's age, gender, height, and weight; Review the patient's past medical history (especially whether there is a history of brittle fractures, whether there is a history of using drugs that affect bone metabolism, etc.).
2. Retrieve the bone density values of the anterior lumbar vertebrae 1 to 4 measured by GE Healthcare Lunar Prodigy dual energy X-ray absorptiometry from the database, and take the average (DXA bone density value). According to the diagnostic criteria of the Diagnosis and Treatment Guidelines for Primary Osteoporosis (2022), determine whether the patient has normal bone mass, decreased bone mass, or osteoporosis.
3. Identify the lumbar spine bone density values (QCT bone density values) measured by the GE Gemstone CTHD750 CT instrument from the database. According to the diagnostic criteria of the Chinese Quantitative CT (QCT) Diagnosis Guidelines for Osteoporosis (2018), determine whether the patient has normal bone mass, decreased bone mass, or osteoporosis.
4. Statistical analysis was conducted on the normal bone density, bone loss, and number of osteoporosis diagnosed by DXA and QCT respectively, in order to explore the differences in the detection rates of osteoporosis between these two monitoring methods. The data was analyzed and processed using SPSS 21.0 statistical software, and the count data was expressed as a rate (%) χ 2-test, P<0.05 indicates statistically significant difference; Explore whether the difference in detection rates between the two is related to factors such as weight; Calculate the detection rates of osteoporosis using two detection methods in patients who have experienced brittle fractures, and preliminarily determine which detection method is more accurate in determining osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and above, regardless of gender
2. The interval between DXA and QCT examinations shall not exceed 3 months.

Exclusion Criteria:

1. Individuals with other metabolic and bone diseases causing focal bone destruction of the vertebral body
2. Incomplete key information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 72 adult patients who underwent lumbar spine anteroposterior DXA and QCT examinations at Qianfoshan Hospital in Shandong Province from January 2019 to December 2022 were selected, with an interval of no more than 3 months between the two examinations for the same patient.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the difference in detection rates of osteoporosis between dual energy X-ray and quantitative CT | January 2019 to December 2022
  Statistical analysis was conducted on the normal bone density, bone loss, and number of osteoporosis diagnosed by DXA and QCT respectively, in order to explore the differences in the detection rates of osteoporosis between these two monitoring methods. The data was analyzed and processed using SPSS 21.0 statistical software, and the count data was expressed as a rate (%) χ 2-test, P<0.05 indicates statistically significant difference; Explore whether the difference in detection rates between the two is related to factors such as weight; Calculate the detection rates of osteoporosis using two detection methods in patients who have experienced brittle fractures, and preliminarily determine which detection method is more accurate in determining osteoporosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No